CLINICAL TRIAL: NCT01871948
Title: Effective Communication for Preventing and Responding to Oncology Adverse Events
Acronym: CanComm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kathleen Mazor, Associate Professor of Medicine, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1184; P20CA137219 (NIH)
Record Dates: First submitted 2013-05-22; First posted 2013-06-07 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient survey at 2 points in time (No Intervention): Randomly assigned patients attending cancer clinics at Washington or Georgia sites during February 2013 to August 2013 will be presented with or mailed a survey about cancer communication approximately 2 weeks later and a follow-up survey approximately 3 months later.
- "WeWant to Know" campaign, patient survey at 2 time points (Experimental): Randomly assigned patients attending cancer clinics at Washington or Georgia sites during February 2013 to August 2013 will be presented with or mailed a survey about cancer communication approximately 2 weeks later and a follow-up survey approximately 3 months later. Additionally, this group will also receive a follow-up phone call approximately 4 weeks after baseline survey.
  Interventions: Other: "We Want to Know" campaign, Patient survey at 2 time points

INTERVENTIONS:
Other: "We Want to Know" campaign, Patient survey at 2 time points — Randomly assigned patients attending cancer clinics at Washington or Georgia sites during February 2013 to August 2013 will be presented with or mailed a survey about cancer communication approximately 2 weeks later and a follow-up survey approximately 3 months later. Additionally, this group will also receive a follow-up phone call approximately 4 weeks after baseline survey.
  Arms: "WeWant to Know" campaign, patient survey at 2 time points

SUMMARY:
Cancer patients often experience problems in their care, many of which are caused by communication breakdowns. Some communication breakdowns lead to adverse events and even harmful errors. Deficiencies in provider-patient communication can compound patients' distress, lower the quality of care, and disrupt patient-provider relationships. There is little research on patients' and providers' experiences of the communication breakdowns that precipitate adverse events and errors, or on effective responses to these events. Because of this, cancer providers are unsure how to communicate with patients in these difficult situations. The goal of the proposed study is to improve patient-centered communication around adverse events and errors in cancer care. Our specific aims are: 1) To describe patients' experiences with communication around adverse events and errors in cancer care, 2) To describe providers' experiences and practices with communication around adverse events and errors in cancer care, 3) To develop practical recommendations, provider training materials and patient educational materials for improving communication around adverse events and errors in cancer care, 4) To disseminate the recommendations and materials through three health plans, and 5) To conduct a preliminary evaluation of the perceived usefulness and impact of the materials. The investigators will first conduct interviews with breast and colorectal cancer patients who have experienced adverse events or errors at 3 Cancer Research Network (CRN) health plans (Atlanta, Georgia; Seattle, Washington and Worcester, Massachusetts). The interviews will focus on instances where patients believe that better communication might have prevented an adverse event or error, or mitigated the event's impact. Next the investigators will conduct focus groups to understand providers' attitudes and experiences with these communication dilemmas, and use simulations to describe providers' communication practices. Finally, the investigators will interview health plan leaders to identify the systems factors that influence communication with patients around adverse events and errors. These perspectives will be synthesized to create patient and provider educational material for improving communication. Three advisory panels: a Patient Advisory Panel, a Health Plan Advisory Panel and a Dissemination Advisory Panel (including all 14 CRN health plans) will help create and disseminate these educational interventions. Dissemination will occur at the three core clinical sites. The investigators use patient and provider surveys to evaluate the educational materials' impact. This evaluation will provide the evidence-base to refine the study products before widespread dissemination throughout the CRN and beyond. The project will have the advantage of the CRN infrastructure, the CRN Clinical Communication Research Center, and is led by nationally recognized communication researchers.

ELIGIBILITY:
Inclusion Criteria:

* Cancer survivors
* 21 to 80 years of age
* Able to communicate in English
* have adequate hearing
* no cognitive impairments

Exclusion Criteria:

-Any non-melanoma skin cancer, Breast cancer in situ, Cervical intraepithelial neoplasia (CIN): types I, II, III, Stage I colon cancer, Stage IV cancer, Recurrent cancer or second primary

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2008-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Calculate differences in satisfaction with cancer care communication, using a summary score from patient surveys, between intervention and control groups. | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Mazor, EdD, Principal Investigator — University of Massachusetts, Worcester; Thomas H Gallagher, MD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Kaiser Permanente Georgia, Atlanta, Georgia
  - Group Health, Seattle, Washington